CLINICAL TRIAL: NCT03331861
Title: Metformin in Heart Failure Without Diabetes
Acronym: Met-HeFT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Barry Fine, Assistant Professor of Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AAAR5389
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin (Experimental): Metformin for 6 months
  Interventions: Drug: Metformin hydrochloride
- Placebo (Placebo Comparator): Matched placebo for 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin hydrochloride — Metformin starting at 500mg twice a day and increasing to 1000mg twice a day for a total of 6 months
  Other Names: Metformin
  Arms: Metformin
Drug: Placebo — Similar dosing regime as active comparator
  Other Names: Placebo Tablet
  Arms: Placebo

SUMMARY:
A pilot clinical research study that will assess the use of the medication metformin for heart failure in patients who are not diabetic and have no evidence of insulin resistance.

DETAILED DESCRIPTION:
Patients (n=50) will received either the study drug metformin or placebo for 4 months. During the study, the patients will undergo extensive testing that will include symptom assessment, exercise capacity, echocardiography, cardiac PET imaging and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Age >18yrs old
* Patients with chronic heart failure (defined as >6 months duration) uptitrated to recommended or maximally tolerated dose of ACE-I/ARB (unless contraindicated) and beta-blocker (unless contraindicated). If indicated, an aldosterone receptor antagonist should be given (unless contraindicated). An ICD and/or CRT should be implanted, if indicated. Patients with a CRT device should be treated for > 3 months.
* Reduced ejection fraction defined as LVEF ≤ 35%
* NYHA-class II or III with stable symptoms for at least the past 3 months
* Renal Function by eGFR ≥ 45 ml/min (MDRD equation) in accordance with FDA guidance on metformin use in CKD(24)
* Non-insulin resistant defined as a fasting insulin resistance index, or HOMA-IR of <2.7.
* Non-diabetic defined as a HgbA1c <6.0

Exclusion Criteria:

* Any oral or injectable hypoglycemic therapy (e.g. insulin, sulfonylureas)
* Known allergy to metformin or major side effects to metformin treatment
* Concomitant use of a carbonic anhydrase inhibitor (such as acetazolamide or topirafmate)
* Heart Failure Hospitalizations in the past 3 months (primary diagnosis on admission is heart failure)
* Acute myocardial infarction, unstable angina or revascularization with prior 3 months at the time of randomization
* Planned coronary revascularization, heart surgery, CRT implantation or other intervention during the study period that would potentially affect the function of the heart
* Significant, uncorrected primary cardiac valve disease, specifically severely stenotic or regurgitant mitral or aortic valves
* Cardiac arrest or life threatening ventricular arrhythmias within the last 3 months (unless treated with an ICD)
* Atrial fibrillation with poorly controlled ventricular rate at rest (> 110 beats/min)
* Hypertrophic or restrictive cardiomyopathy, infiltrative or storage myocardial disease, active myocarditis, or pericardial disease.
* Planned major surgery within the study period
* Female patients who are pregnant, nursing, or of childbearing potential while not practicing effective chemical contraceptive methods (i.e. oral, implanted, injectable, or transdermal contraceptive hormones; intrauterine device)
* Current abuse of alcohol or drugs
* Life-expectancy of less than 1 year due to co-existing morbid illness
* Liver disease with ALT or AST >3 times upper normal limit (it is possible to repeat this measurement once within a month)
* Advanced lung disease such as COPD
* Significant comorbidity or issue that makes the patient unsuitable for participation as judged by the investigator
* Participation in another study involving long-term medical intervention (participation in device studies is allowed)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Fine, MD, Principal Investigator — Columbia University
Locations (1):
- New York Hospital - Columbia University Irving Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 out of 6 participants screen failed and no further information was collected or analyzed.
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Minute Ventilation to Carbon Dioxide Production (VE/VCO2) Slope
Description: The VO2 change outcomes will be assessed for normality using standard visual assessments (Q-Q plots and histograms) and statistical tests (Kolmogorov-Smirnov). VE/VCO2 slope change will be calculated.
Time Frame: Baseline and 6 months
Population: Study was terminated early; data was not collected due to low enrollment, thus cannot be analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Visual Analog Scale (VAS) Score
Description: Dyspnea Assessment. 100mm line scale ranging from 0 (worse imaginable breathing) to 100 (best imaginable breathing).
Time Frame: Baseline and 6 months
Population: Study was terminated early; data was not collected due to low enrollment, thus cannot be analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Minnesota LIVING WITH HEART FAILURE Questionnaire (MLHFQ) Score
Description: A validated patient-oriented measure of the adverse effects of heart failure on a patient's life. The questionnaire is comprised of 21 questions around several physical, emotional and socioeconomic ways heart failure can adversely affect a patient's life. After receiving brief standardized instructions, the patient marks a 0 (zero) to 5 (five) scale to indicate the extent to which each itemized adversity of heart failure has prevented the patient from living as they wanted to live during the past 4 weeks. The questionnaire is simply scored by summation of all 21 responses.
Time Frame: Baseline, 6 months
Population: Study was terminated early; data was not collected due to low enrollment, thus cannot be analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Peak Myocardial Oxygen Consumption (VO2)
Description: Oxygen consumption (VO2) (ml/min) will be measured on a breath by breath basis. Peak VO2 will be computed using standard methods.
Time Frame: Baseline, 6 months
Population: Study was terminated early; data was not collected due to low enrollment, thus cannot be analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Heart Failure Hospitalizations
Description: The number of hospitalizations recorded during the study will be tallied.
Time Frame: Up to 6 months
Population: Study was terminated early; data was not collected due to low enrollment, thus cannot be analyzed.
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Study was terminated early, data was unblinded but not analyzed due to low enrollment and lack of statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT03331861/Prot_SAP_000.pdf